CLINICAL TRIAL: NCT02093650
Title: Black Cohosh Extract for the Treatment of Moderate to Severe Menopausal Symptoms: a Randomized-placebo Controlled Trial
Brief Title: Black Cohosh Extract for Treatment of Moderate to Severe Menopausal Symptoms
Acronym: BCOMS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Patsama Vichinsartvichai, MD., Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 081/56; TCTR20140318001 (Registry Identifier: Thai Clinical Trials Registry)
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Menopause; Quality of Life
Keywords: Menopausal symptoms; menopause related quality of life; black cohosh; cimicifuga racemosa; MENQOL; Kupperman index; KI; liver function tests
MeSH Terms: interventions — black cohosh root extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Black cohosh extract (Active Comparator): black cohosh extract 80 mg daily
  Interventions: Drug: black cohosh extract
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: black cohosh extract — Black cohosh extract 80 mg
  Other Names: Femosa
  Arms: Black cohosh extract
Drug: Placebo — Soy bean oil
  Arms: Placebo

SUMMARY:
Compare the treatment efficacy of black cohosh extract 80 mg daily and placebo for moderate to severe menopausal symptoms

DETAILED DESCRIPTION:
Compare the treatment efficacy of black cohosh extract 80 mg/day an placebo for moderate to severe menopausal symptoms with Kupperman menopausal index and MENQOL

ELIGIBILITY:
Inclusion Criteria:

* Age at least 40 years
* Peri or post menopause
* Moderate to severe menopausal symptoms (Kupperman index at least 20)

Exclusion Criteria:

* Use hormonal treatment or other treatments within 4 weeks
* Use atorvastatin azathioprine or cyclosporin within 4 weeks
* BMI at least 30 kg m2
* Allergic to drug or components
* Liver disease or abnormal liver function test
* Psychiatric disease
* Alcoholic or drug abuse
* Vegetarian

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The changes in Kupperman Index | baseline, week 4, week 8 and week 12
  Kupperman index questionnaire at baseline, 4, 8 and 12 weeks

SECONDARY OUTCOMES:
A change in MENQOL | baseline and week 12
  MENQOL questionnaire measurement at baseline and 12 weeks
The changes in daily hot flushes frequency | baseline, week 4, week 8 and week 12
  Daily hot flushes frequency over 12 weeks treatment
Global satisfaction | week 12
  Overall patient satisfaction 0 - 10 scale
A change in liver function test | baseline and week 12
  Changes in liver function test from baseline and 12 weeks
adverse events | week 4, week 8 and week 12
  frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Patsama Vichinsartvichai, MD, Principal Investigator — Faculty of Medicine Vajira Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine Vajira Hospital, Navamindradhiraj University, Dusit, Bangkok, Thailand